CLINICAL TRIAL: NCT06101667
Title: Efficacy and Safety of Endovascular Recanalization for Acute Basilar Artery Occlusion With Extended Time Window -- A Multicenter, Prospective, Open-label, Blind Endpoint, Randomized Controlled Trial（ANGEL-BAO）
Brief Title: Efficacy and Safety of Endovascular Recanalization for Acute Basilar Artery Occlusion With Extended Time Window (ANGEL-BAO)
Acronym: ANGEL-BAO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Feng Gao, Vice-Director of Interventional Neuroradiology, Department of Neurology, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HX-A-2023021
Record Dates: First submitted 2023-10-15; First posted 2023-10-26 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Acute Ischemic Stroke; Basilar Artery Occlusion
Keywords: Acute Ischemic Stroke; Basilar Artery Occlusion; Extended Time Window; Endovascular Treatment
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Best medical management (Active Comparator): Patients randomly assigned to the control group should receive the best medical management according to the guidelines.
  Interventions: Drug: Best medical management
- Endovascular treatment (Experimental): Stent retrievers, thromboaspiration, balloon angioplasty, stent deployment, intra-arterial thrombolysis (Recombinant tissue plasminogen activator (rt-PA) or urokinase), or the various combinations of these approaches.
  Interventions: Procedure: Endovascular treatment

INTERVENTIONS:
Drug: Best medical management — Best medical management included assessment of vital signs and neurological deficits,airway protection respiratory support,circulation;blood pressure monitoring;nutritional support;complication control;symptomatic treatment;laboratory and imaging examinations;etiological analysis and evaluation; anti platelet（e.g. aspirin,adenosine diphosphate (ADP) receptor inhibitors,Adenosine reuptake inhibitors,Glycoprotein platelet inhibitors）；anticoagulation(e.g. warfarin, rivaroxaban,dabigatran,apixaban,edoxaban)；lipid lowering(e.g. Statins,Fibrates）；control of blood pressure(e.g. Thiazide diuretics,Potassium-sparing,Loop diuretic,Beta-blockers,Angiotensin II receptor blockers,Calcium channel blockers,Alpha blockers,Central alpha-2 receptor agonists);control of blood glucose(e.g. SULFONYLUREAS (SFUs),GLINIDES,BIGUANIDES,ALPHA-GLUCOSIDASE INHIBITORS: STARCH BLOCKERS,THIAZOLIDINEDIONES,GLP-1 ANALOGS,DPP-4 INHIBITORS,SGLT2 inhibitors); control of other risk factors
  Arms: Best medical management
Procedure: Endovascular treatment — The strategies that were used for endovascular treatment included :stent retrievers (e.g., Solitaire® [Medtronic, USA], Trevo® [Stryker, USA], EMBOTRAP® [Johnson & Johnson, USA], Captor® [HeartCare, China] and other stent-retriever systems) thromboaspiration (e.g., Penumbra® [Penumbra, USA], Afentta® [HeMo, China] and other aspiration systems)) balloon angioplasty (e.g., Gateway® [Stryker, USA], Neuro RX® [SinoMed, China], FocuStar® [HeMo, China] and other intracranial balloon catheter systems) stent deployment (e.g., Wingspan® [Stryker, USA], Apollo® [MircoPort, China], Enterprise® [Johnson & Johnson, USA], Neuroform EZ® [Stryker, USA] and other Intracranial stent systems)) intraarterial thrombolysis (with alteplase or urokinase) combinations of above approaches that were left to the discretion of the treating team
  Arms: Endovascular treatment

SUMMARY:
The aim of this study is to assess the efficacy and safety of endovascular treatment versus medical management in patients with acute basilar artery occlusion with extended time window of 24-72 hours from onset.

DETAILED DESCRIPTION:
The ANGEL-BAO is a multicentered, prospective, randomized, open-label, blinded end-point clinical trial. A total of 224 patients with acute basilar artery occlusion with extended time window of 24-72 hours from onset will be enrolled. Patients fulfilling all of the inclusion criteria and none of the exclusion criteria will be randomized 1:1 into two groups (endovascular treatment or medical management) after offering informed content.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years
2. Acute basilar artery occlusion confirmed by CTA, MRA, or DSA
3. Pre-stroke mRS of 0-2
4. NIHSS score ≥ 10 before randomization
5. Time interval from symptom onset (or last known well) to randomization within 24-72 hours
6. Diffusion-weighted imaging(DWI)-based pc-ASPECTS ≥ 6 and Pons-Midbrain Index (PMI) ≤3
7. Time from completion of DWI imaging to randomization is ≤3 hours
8. Each patient or their legal representative must provide written informed consent before enrolment

Exclusion Criteria:

1. Any sign of intracranial hemorrhage (except microbleeds) on brain imaging prior to randomization
2. Complete cerebellar infarct with significant mass effect, or bilateral thalamic infarction as evidenced by baseline neuroimaging
3. CT or MRI evidence of intracranial tumor (except small meningioma and cerebral aneurysm < 3mm in diameter)
4. Known or highly suspected chronic occlusion of basilar artery
5. History of contraindication for contrast medium (except mild rash)
6. Current pregnant or breast-feeding
7. Known to have dementia or psychiatric disease unable to complete neurological assessment and follow-up
8. Life expectancy is less than 3 months
9. Enrolled in another drug or device trial or expected to participate in another drug or device treatment trial within the following 3 months.
10. Any other condition (in the opinion of the site investigator) that inappropriate to participate this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rate of modified Rankin scale 0-3 at 90 (±14) days after randomization | 90±14 days after randomization
  The modified Rankin scale (mRS) ranged from 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death.

SECONDARY OUTCOMES:
MRS score as an ordinal scale at 90 (±14) days after randomization | 90±14 days after randomization
  The modified Rankin scale (mRS) ranged from 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death.
Rate of mRS 0-2 at 90 (±14) days after randomization | 90±14 days after randomization
  The modified Rankin scale (mRS) ranged from 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death.
National Institutes of Health Stroke Scale (NIHSS) score at 24 hours after randomization | 24 hours after randomization
  The National Institute of Health Stroke Scale（NIHSS） ranged from 0 to 42, with higher scores indicating greater neurologic deficits.
NIHSS score at 7 days after randomization or discharge (whichever came first) | 7 days after randomization or at discharge
  The National Institute of Health Stroke Scale（NIHSS） ranged from 0 to 42, with higher scores indicating greater neurologic deficits.
Functional health status and quality of life (EuroQol Five Dimensions) at 90 (±14) days after randomization | 90±14 days after randomization
  EuroQol Five Dimensions (EQ-5D) is a standardized instrument for measuring the general health status. Rated level can be coded as a number 1, 2, 3, 4 or 5, which indicates having no problems for 1, having some problems for 2, having moderate problems for 3, having serious problems for 4 and having extreme problems for 5.
Proportion of basilar artery recanalization at 18-36 hours after randomization (confirmed by CTA or MRA) | 18-36 hours after randomization
  Basilar artery recanalization is defined as grade 2-3 of arterial occlusive lesion (AOL) scale.
  The AOL Score was defined as: 0=no recanalization of the primary occlusion, 1=incomplete or partial recanalization of the primary occlusion with no distal flow, 2=incomplete or partial recanalization of the primary occlusion with distal flow, or 3=complete recanalization of the primary occlusion with distal flow.

OTHER OUTCOMES:
Rate of any Symptomatic intracranial hemorrhage (SICH) defined as the Heidelberg classification within 18-36 hours of randomization | 18-36 hours after randomization
  Heidelberg standard was defined as new intracranial hemorrhage detected by brain imaging associated with any of the item below: 4 points total NIHSS at the time of diagnosis compared to immediately before worsening. 2 point in one NIHSS category. Leading to intubation/hemicraniectomy/ventricular drainage placement or other major medical/surgical intervention. Absence of alternative explanation for deterioration.
Rate of any Any intracranial hemorrhage identified by CT or MRI imaging within 18-36 hours after randomization | Any intracranial hemorrhage identified by CT or MRI imaging within 18-36 hours
  Any intracranial hemorrhage identified by CT or MRI imaging within 18-36 hours
All cause of mortality within 7 days after randomization | 7 days after randomization
  All cause of mortality within 7 days after randomization
All cause of mortality within 90 (±14) days after randomization | 90±14 days after randomization
  All cause of mortality within 90 (±14) days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Feng Gao, MD, Principal Investigator — Beijing Tiantan Hospital, Capital Medical Univerity; Zhongrong Miao, PhD, Principal Investigator — Beijing Tiantan Hospital, Capital Medical Univerity
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No